CLINICAL TRIAL: NCT02319161
Title: Comparison of Calcium-channel Blockers and Beta Blockers in Tourniquet-induced Hypertension During Intravenous Regional Anesthesia
Brief Title: Comparison of Calcium Channel Blockers and Beta Blockers on Tourniquet-induced Hypertension During Intravenous Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Specialist, Ankara University
Other Study IDs: 04-130-14
Record Dates: First submitted 2014-12-13; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
Keywords: intravenous regional anesthesia
MeSH Terms: conditions — Hypertension | interventions — Calcium Channel Blockers; Adrenergic beta-Antagonists; esmolol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: Group I: the patients with systolic blood pressure above to 150 mmHg following tourniquet inflation and in which bolus dose of calcium channel blocker 10 mg was administered by intravenous route.
  Interventions: Drug: Calcium channel blocker and beta blocker
- Group II: Group II: the patients with systolic blood pressure above to 150 mmHg following tourniquet inflation and in which bolus dose of beta blocker 0.5mg/kg was administered by intravenous route
  Interventions: Drug: Calcium channel blocker and beta blocker

INTERVENTIONS:
Drug: Calcium channel blocker and beta blocker — The patients in which systolic blood pressure increased to 150 mmHg and above following tourniquet inflation and in which a bolus dose of calcium channel blocker 10 mg (Diltizem, Mustafa Nevzat İlaç Sanayi Aş) (Group I) or beta blocker 0.5mg/kg (Brevibloc, Eczacıbaşı İlaç Sanayi Aş) (Group II) were administered intravenously constituted the study groups.
  Other Names: Diltizem , Brevibloc

SUMMARY:
The investigators aimed to investigate the efficacy of calcium channel blockers and beta blockers for controlling tourniquet induced blood pressure increase in patients undergoing carpal tunnel operations with IVRA. For this purpose files of patients undergoing operation under IVRA were retrospectively examined in terms of demographical and hemodynamic variables.

DETAILED DESCRIPTION:
After approval of the University Research Ethics Committee, the files of patients who have been operated under intravenous regional anesthesia (IVRA) in orthopedics clinics between January 2009 and January 2010 were retrospectively investigated. A total of 312 patients, 164 patients with carpal tunnel syndrome and 148 patients with trigger finger have been operated under IVRA. Out of 164 patients who have been operated due to carpal tunnel syndrome, 50 patients in which either calcium channel blockers or beta blockers were used for treatment of critical blood pressure increase after tourniquet inflation and in which whole data were obtained, were included to the study.The patients with systolic blood pressure above to 150 mmHg following tourniquet inflation and in which bolus dose of diltiazem 10 mg (Group I) or calcium channel blocker 0.5mg/kg (Group II) have been administered by intravenous route constituted the study groups. Demographical characteristics and hemodynamic parameters were recorded from the patient files.

ELIGIBILITY:
Inclusion Criteria:

Patients operated due to carpal tunnel syndrome under intravenous regional anesthesia betweem January 2009 and January 2010.

Exclusion Criteria:

The patients that the files could not be reached

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The files of patients who were operated on under intravenous regional anesthesia (IVRA) in orthopedics clinics between January 2009 and January 2010 were retrospectively investigated. A total of 312 patients, 164 patients with carpal tunnel syndrome and 148 patients with trigger finger were operated on under IVRA. Out of 164 patients who were operated on due to carpal tunnel syndrome, 50 patients in which either calcium channel blockers or beta blockers were used for treatment of critical blood pressure increase after tourniquet inflation and in which whole data were obtained, were included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Decrease in blood pressure | 2 hours

SECONDARY OUTCOMES:
Decrease in pain | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: K. Sanem Çakar Turhan, Specialist, Principal Investigator — Ankara University Medical Faculty